CLINICAL TRIAL: NCT01289184
Title: Air Quality Monitoring and Health Surveillance of Workers in the Photocopier Units
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Avinashilingam Deemed University (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Dr.G.P.JEYANTHI, PROFESSOR, DEPARTMENT OF BIOCHEMISTRY, BIOTECHNOLOGY AND BIOINFORMATICS, AVINASHILINGAM DEEMED UNIVERSITY FOR WOMEN,COIMBATORE 641043
Other Study IDs: AIR QUALITY IN PHOTOCOPY UNITS
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-01

CONDITIONS: Occupational Exposure
Keywords: Occupational Health Hazards; Air Pollution; Photocopiers; Other Specified Personal Exposures; History Presenting Hazards to Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- control
- exposure 2-3 years
- exposure 3-5 years
- exposure 5-10 years
- exposure >15 years

SUMMARY:
To monitor air quality in selected photocopier units and to assess the health status of workers who are exposed to emissions from photocopiers.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 years of exposure to photocopiers

Exclusion Criteria:

* any clinical abnormality

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: At least two years of working experience in photocopier units
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Avinashilingam Deemed University For Women, Coimbatore, Tamil Nadu, India